CLINICAL TRIAL: NCT02597218
Title: Incidence of Venous Thromboembolic Disease and Portal Vein Thrombosis After Hepatectomy in a High-volume Center. A Cohort Study.
Brief Title: Incidence of Venous Thromboembolic Disease and Portal Vein Thrombosis After Hepatectomy. A Cohort Study.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, Diego Hernan Giunta, MD, MD, Hospital Italiano de Buenos Aires
Other Study IDs: 2611
Record Dates: First submitted 2015-11-03; First posted 2015-11-05 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Pulmonary Embolism; Venous Thrombosis; Portal Thrombosis
Keywords: Hepatectomy; Prophylaxis
MeSH Terms: conditions — Pulmonary Embolism; Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients following hepatectomy: Patients following hepatectomy of any type, any gender. Roughly, we will describe: type of resection, presence of cancer,use of mechanical/pharmacological prophylaxis, major/minor bleedings ocurring during observation period.
  Outcomes: Venous thromboembolism (VTE)[deep vein thrombosis (DVT) and pulmonary embolism (PE)] and portal thrombosis (PT).

SUMMARY:
Observational. Retrospective cohort.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE) is a disease that includes both deep vein thrombosis (DVT) and pulmonary embolism (PE). It is a common, potentially lethal disorder that can occur among postoperative patients. Liver surgery implies a prothrombotic state, as a result of an alteration of the equilibrium between synthesis and use of pro and anti coagulant factors after a parenquimal resection. The use of antithrombotic prophylaxis following surgery is not standarized, and current practices vary depending on the attendant surgeon's particular experience or hospital's customs and habits.

In published research, postoperative patients have been studied as a whole so far. There is little evidence regarding patients undergoing hepatectomy. Furthermore, the use and need of extended prophylaxis remains unexplored in this group of patients.

The objetives of the following study are:

* To estimate the incidence of symptomatic venous thromboembolism (VTE) [deep vein thrombosis (DVT), pulmonary embolism (PE) and fatal PE] in a third level center in patients undergoing any hepatectomy within 90 days after surgery.
* To estimate the incidence of portal thrombosis (PT) in a third level center in patients undergoing any hepatectomy within 90 days after surgery.
* To identify and describe factors associated to the development of VTE in patients following hepatectomy.
* To identify and describe factors associated to the development of PT in patients following hepatectomy.
* To describe major bleedings or minor but clinically relevant bleedings during the period in which those patients received chemical thromboprophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old.
* Following hepatic surgery.

Exclusion Criteria:

* Living donor
* Venous thromboembolism within 6 months previous to surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years following hepatectomy of any kind for oncologic/non-oncologic disease between 04/09/2012 and 08/28/2015 were enrolled. Follow-up concluded 90 days after surgery or at occurence of event (Venous thromboembolism / portal thrombosis / death).
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2015-10; Primary Completion 2019-10 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Venous thromboembolism (VTE) | 90 days following surgery
  Includes deep vein thrombosis (DVT) and pulmonary embolism (PE)

SECONDARY OUTCOMES:
Portal Thrombosis (PT) | 90 days following surgery
  Portal thrombosis
Minor bleeding | 90 days following surgery
  Any bleeding that doesn't fulfill "major bleeding" criteria.
Major bleeding | 90 days following surgery
  Any bleeding causing: death, serious threat to life, requirement of active medical intervention, 2 or more red blood cell units transfusion, localized in retroperitoneum, intracraneal or intraocular

CONTACTS AND LOCATIONS:
Overall Officials: Martín de Santibañes, Dr, Study Director — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Capital Federal, Buenos Aires, Argentina

REFERENCES:
- [Background] Rasmussen MS. Preventing thromboembolic complications in cancer patients after surgery: a role for prolonged thromboprophylaxis. Cancer Treat Rev. 2002 Jun;28(3):141-4. doi: 10.1016/s0305-7372(02)00043-9. PMID 12234565
- [Background] Ejaz A, Spolverato G, Kim Y, Lucas DL, Lau B, Weiss M, Johnston FM, Kheng M, Hirose K, Wolfgang CL, Haut E, Pawlik TM. Defining incidence and risk factors of venous thromboemolism after hepatectomy. J Gastrointest Surg. 2014 Jun;18(6):1116-24. doi: 10.1007/s11605-013-2432-x. Epub 2013 Dec 13. PMID 24337986
- [Background] Caprini JA, Arcelus JI, Hasty JH, Tamhane AC, Fabrega F. Clinical assessment of venous thromboembolic risk in surgical patients. Semin Thromb Hemost. 1991;17 Suppl 3:304-12. PMID 1754886
- [Background] Collins R, Scrimgeour A, Yusuf S, Peto R. Reduction in fatal pulmonary embolism and venous thrombosis by perioperative administration of subcutaneous heparin. Overview of results of randomized trials in general, orthopedic, and urologic surgery. N Engl J Med. 1988 May 5;318(18):1162-73. doi: 10.1056/NEJM198805053181805. No abstract available. PMID 3283548
- [Background] Prevention of fatal postoperative pulmonary embolism by low doses of heparin. An international multicentre trial. Lancet. 1975 Jul 12;2(7924):45-51. PMID 49649
- [Background] Kiil J, Kiil J, Axelsen F, Andersen D. Prophylaxis against postoperative pulmonary embolism and deep-vein thrombosis by low-dose heparin. Lancet. 1978 May 27;1(8074):1115-6. doi: 10.1016/s0140-6736(78)90297-0. PMID 77413
- [Background] Pezzuoli G, Neri Serneri GG, Settembrini P, Coggi G, Olivari N, Buzzetti G, Chierichetti S, Scotti A, Scatigna M, Carnovali M. Prophylaxis of fatal pulmonary embolism in general surgery using low-molecular weight heparin Cy 216: a multicentre, double-blind, randomized, controlled, clinical trial versus placebo (STEP). STEP-Study Group. Int Surg. 1989 Oct-Dec;74(4):205-10. PMID 2560470
- [Background] Mismetti P, Laporte S, Darmon JY, Buchmuller A, Decousus H. Meta-analysis of low molecular weight heparin in the prevention of venous thromboembolism in general surgery. Br J Surg. 2001 Jul;88(7):913-30. doi: 10.1046/j.0007-1323.2001.01800.x. PMID 11442521
- [Background] Gould MK, Garcia DA, Wren SM, Karanicolas PJ, Arcelus JI, Heit JA, Samama CM. Prevention of VTE in nonorthopedic surgical patients: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e227S-e277S. doi: 10.1378/chest.11-2297. PMID 22315263
- [Background] Lyman GH, Khorana AA, Kuderer NM, Lee AY, Arcelus JI, Balaban EP, Clarke JM, Flowers CR, Francis CW, Gates LE, Kakkar AK, Key NS, Levine MN, Liebman HA, Tempero MA, Wong SL, Prestrud AA, Falanga A; American Society of Clinical Oncology Clinical Practice. Venous thromboembolism prophylaxis and treatment in patients with cancer: American Society of Clinical Oncology clinical practice guideline update. J Clin Oncol. 2013 Jun 10;31(17):2189-204. doi: 10.1200/JCO.2013.49.1118. Epub 2013 May 13. PMID 23669224
- [Background] Barton JS, Riha GM, Differding JA, Underwood SJ, Curren JL, Sheppard BC, Pommier RF, Orloff SL, Schreiber MA, Billingsley KG. Coagulopathy after a liver resection: is it over diagnosed and over treated? HPB (Oxford). 2013 Nov;15(11):865-71. doi: 10.1111/hpb.12051. Epub 2013 Jan 29. PMID 23458574
- [Background] Bezeaud A, Denninger MH, Dondero F, Saada V, Venisse L, Huisse MG, Belghiti J, Guillin MC. Hypercoagulability after partial liver resection. Thromb Haemost. 2007 Dec;98(6):1252-6. PMID 18064322
- [Background] Tzeng CW, Katz MH, Fleming JB, Pisters PW, Lee JE, Abdalla EK, Curley SA, Vauthey JN, Aloia TA. Risk of venous thromboembolism outweighs post-hepatectomy bleeding complications: analysis of 5651 National Surgical Quality Improvement Program patients. HPB (Oxford). 2012 Aug;14(8):506-13. doi: 10.1111/j.1477-2574.2012.00479.x. Epub 2012 May 15. PMID 22762398
- [Background] Smyrniotis V, Farantos C, Kostopanagiotou G, Arkadopoulos N. Vascular control during hepatectomy: review of methods and results. World J Surg. 2005 Nov;29(11):1384-96. doi: 10.1007/s00268-005-0025-x. PMID 16222453
- [Background] Yoshiya S, Shirabe K, Nakagawara H, Soejima Y, Yoshizumi T, Ikegami T, Yamashita Y, Harimoto N, Nishie A, Yamanaka T, Maehara Y. Portal vein thrombosis after hepatectomy. World J Surg. 2014 Jun;38(6):1491-7. doi: 10.1007/s00268-013-2440-8. PMID 24407940
- [Background] Weiss MJ, Kim Y, Ejaz A, Spolverato G, Haut ER, Hirose K, Wolfgang CL, Choti MA, Pawlik TM. Venous thromboembolic prophylaxis after a hepatic resection: patterns of care among liver surgeons. HPB (Oxford). 2014 Oct;16(10):892-8. doi: 10.1111/hpb.12278. Epub 2014 May 28. PMID 24888461
- [Background] Tzeng CW, Curley SA, Vauthey JN, Aloia TA. Distinct predictors of pre- versus post-discharge venous thromboembolism after hepatectomy: analysis of 7621 NSQIP patients. HPB (Oxford). 2013 Oct;15(10):773-80. doi: 10.1111/hpb.12130. Epub 2013 Jul 22. PMID 23869577
- [Background] Agnelli G, Bolis G, Capussotti L, Scarpa RM, Tonelli F, Bonizzoni E, Moia M, Parazzini F, Rossi R, Sonaglia F, Valarani B, Bianchini C, Gussoni G. A clinical outcome-based prospective study on venous thromboembolism after cancer surgery: the @RISTOS project. Ann Surg. 2006 Jan;243(1):89-95. doi: 10.1097/01.sla.0000193959.44677.48. PMID 16371741
- [Background] Bergqvist D, Agnelli G, Cohen AT, Eldor A, Nilsson PE, Le Moigne-Amrani A, Dietrich-Neto F; ENOXACAN II Investigators. Duration of prophylaxis against venous thromboembolism with enoxaparin after surgery for cancer. N Engl J Med. 2002 Mar 28;346(13):975-80. doi: 10.1056/NEJMoa012385. PMID 11919306
- [Background] Posadas-Martinez ML, Vazquez FJ, Giunta DH, Waisman GD, de Quiros FG, Gandara E. Performance of the Wells score in patients with suspected pulmonary embolism during hospitalization: a delayed-type cross sectional study in a community hospital. Thromb Res. 2014 Feb;133(2):177-81. doi: 10.1016/j.thromres.2013.11.018. Epub 2013 Nov 25. PMID 24342535